CLINICAL TRIAL: NCT05828953
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Trial of Anlotinib Capsules for the Treatment of Idiopathic Pulmonary Fibrosis (IPF)/Progressive Fibrosis-interstitial Lung Disease (PF-ILDs)
Brief Title: Anlotinib Capsules in the Treatment for IPF/PF-ILDs
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xiaoying Huang, Vice-president of First Affiliated Hospital of Wenzhou Medical University, First Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ky2021-128-01
Record Dates: First submitted 2023-03-27; First posted 2023-04-25 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Interstitial Lung Diseases
Keywords: Idiopathic pulmonary fibrosis(IPF); Progressive fibrosis-interstitial lung disease(PF-ILDs); Anlotinib
MeSH Terms: conditions — Lung Diseases, Interstitial; Idiopathic Pulmonary Fibrosis | interventions — anlotinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anlotinib (Experimental): Experimental: The dosage of Anlotinib is 8mg per dose, once daily, to be taken orally before breakfast.
  Interventions: Drug: Anlotinib
- Placebo, (Placebo Comparator): control group：Placebo, take orally once daily before breakfast
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anlotinib — Drug: Anlotinib The dose of nintedanib hydrochloride is 8mg per dose, taken orally once daily before breakfast. The drug is taken continuously for 2 weeks, followed by a 1-week break, until week 52, disease progression, or the occurrence of intolerable adverse events. If a dose is missed and the next dose is due within 12 hours, it should not be made up.
  Drug: Placebo Placebo, taken orally once daily before breakfast. Taken continuously for 2 weeks, followed by a 1-week break, until week 52, disease progression, or the occurrence of intolerable adverse events. If a dose is missed and the next dose is due within 12 hours, it should not be made up.
  Arms: Anlotinib
Drug: Placebo — Placebo, taken orally once daily before breakfast. Taken continuously for 2 weeks, followed by a 1-week break, until week 52, disease progression, or the occurrence of intolerable adverse events. If a dose is missed and the next dose is due within 12 hours, it should not be made up.
  Arms: Placebo,

SUMMARY:
The use of Anlotinib hydrochloride capsules for the treatment of IPF/PF-ILDs, with FVC as the primary efficacy endpoint to evaluate its effectivenes

DETAILED DESCRIPTION:
Drug: Anlotinib The dose of nintedanib hydrochloride is 8mg per dose, taken orally once daily before breakfast. The drug is taken continuously for 2 weeks, followed by a 1-week break, until week 52, disease progression, or the occurrence of intolerable adverse events. If a dose is missed and the next dose is due within 12 hours, it should not be made up.

Drug: Placebo Placebo, taken orally once daily before breakfast. Taken continuously for 2 weeks, followed by a 1-week break, until week 52, disease progression, or the occurrence of intolerable adverse events. If a dose is missed and the next dose is due within 12 hours, it should not be made up.

FVC stands for forced vital capacity, which is typically the maximum amount of air that can be forcefully exhaled after taking a deep breath as quickly and completely as possible. This measure primarily assesses the ability to exhale as much air as possible in the shortest amount of time, and is used as an indicator of lung function.The change in FVC from baseline at week 52 after administration.

ELIGIBILITY:
Inclusion Criteria:

1. The participants voluntarily joined the study and signed an informed consent form. They showed good compliance throughout the study.
2. The study includes individuals aged 40-85 years old, of any gender, with an expected lifespan of over 1 year.
3. Subjects who meet either of the following two criteria: a. HRCT results confirming IPF diagnosis within the past 5 years and HRCT results within the past 12 months showing a range of parenchymal fibrotic changes between ≥10% and <50%, with less than 25% honeycombing change in the lung, and no other facilitating factors (e.g. asbestos exposure, allergic pneumonia, systemic sclerosis, rheumatoid arthritis) as detailed in Annex 1A. b. PF-ILDs: Patients with characteristics of fibrotic lung disease (see Annex 1B), and at least one of the following diagnostic criteria is met: i. Relative decline in FVC% predicted by ≥10% within 6 months; ii. Relative decline in FVC% predicted by ≥5-10% with worsening respiratory symptoms, or an increase in the degree of fibrosis on chest HRCT; ii. Worsening respiratory symptoms combined with an increase in the degree of fibrosis on chest HRCT;
4. Carbon monoxide diffusion capacity (DLco) (corrected for hemoglobin) between 30% and 80% of predicted value;
5. Force vital capacity (FVC) ≥ 45% predicted;
6. The 6MWT distance is ≥ 150 meters
7. Arterial partial pressure of oxygen (PaO2) ≥ 60 mmHg (measured at sea level atmospheric pressure, at rest, and breathing room air)
8. "Major organ functions are good, and meet the following criteria: a. Standard blood routine examination (not corrected by blood transfusion or hematopoietic growth factor drugs in the past 7 days): hemoglobin (HGB) ≥ 90 g/L; absolute neutrophil count (NEUT) ≥ 1.5 × 10^9/L; platelet count (PLT) ≥ 90 × 10^9/L; b. Biochemical examination should meet the following criteria: total bilirubin (TBL) ≤ 1.5 times the upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; serum creatinine (Cr) ≤ 1.5 × ULN or creatinine clearance rate (Ccr) ≥ 60 ml/min; c. Coagulation function or thyroid function examination should meet the following criteria: prothrombin time (PT), activated partial thromboplastin time (APTT), international normalized ratio (NR) ≤ 1.5 × ULN (not receiving anticoagulation therapy) or stable use of anticoagulants in the 2 weeks before enrollment; d. Thyroid-stimulating hormone (TSH) ≤ ULN after standard treatment; if abnormal, T3 and T4 levels should be investigated and can be enrolled if T3 and T4 levels are normal.

   e. Echocardiography evaluation: Left ventricular ejection fraction (LVEF) ≥50%
9. Female participants of childbearing potential must agree to use contraception (such as intrauterine device, contraceptive pill, or condom) during the study and for 6 months after the end of the study; must have a negative serum pregnancy test within 7 days before study entry and must not be lactating. Male participants must agree to use contraception during the study and for 6 months after the end of the study.

Exclusion Criteria:

1. Patients with acute exacerbation of PF/PF-ILDs.;
2. Multiple factors that affect oral medication (such as dysphagia, chronic diarrhea, and intestinal obstruction)
3. Received major surgical treatment, incisional biopsy, or significant traumatic injury within 28 days prior to the start of the study treatment.
4. Long-standing non-healing wound or fracture.
5. Patients who have experienced thrombotic events, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, and cerebral infarction), deep vein thrombosis, and pulmonary embolism, within the past 6 months, or those with other bleeding tendencies.
6. Subjects with any severe or uncontrolled comorbidities or undergoing immunotherapy, such as:

   1. Blood pressure remains uncontrolled even after antihypertensive therapy (systolic blood pressure ≥150mmHg or diastolic blood pressure ≥100mmHg); 2nd-degree myocardial ischemia or myocardial infarction, arrhythmia (including QTc ≥450ms (men), QTc ≥470ms (women)) or 2nd-degree congestive heart failure (New York Heart Association (NYHA) classification); pulmonary or systemic infections within 4 weeks before enrollment;
   2. Severe pulmonary arterial hypertension (systolic pulmonary artery pressure (SPAP) ≥70mmHg);
   3. Renal failure requiring hemodialysis or peritoneal dialysis;
   4. History of immune deficiency diseases, including HIV-positive or other acquired or congenital immune deficiency diseases, or history of organ transplantation;
   5. Known clinically significant liver disease history, including viral hepatitis, known carriers of hepatitis B virus (HBV) must exclude active HBV infection, i.e., HBV DNA positive (>2500 copies/mL or >500IU/mL, and greater than the upper limit of normal); known hepatitis C virus (HCV) infection and positive HCV RNA (>1×103 copies/mL), or other decompensated liver diseases;
   6. Fasting blood glucose (FBG) >10mmol/L after administration of hypoglycemic drugs (poor blood glucose control patients);
   7. Urine routine test indicates urine protein ≥+, and 24-hour urine protein quantitation is confirmed to be >1.0g.
7. Received high-dose steroids (e.g. prednisone >15mg/kg) within 1 month prior to randomization；
8. Use of immunosuppressants within 1 month prior to randomization after enrollment;
9. Long-term use (>1 week) of drugs such as amiodarone that may cause pulmonary fibrosis prior to enrollment;
10. Received interferon, N-acetylcysteine (>1800mg), or other anti-fibrotic drugs within 1 month prior to randomization
11. Received treatment with nintedanib or pirfenidone for less than 28 days before randomization.
12. Participation in other drug trials within 3 months prior to randomization
13. The researcher considers any ineligible candidates.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
FVC | 52weeks
  FVC stands for forced vital capacity, which is typically the maximum amount of air that can be forcefully exhaled after taking a deep breath as quickly and completely as possible. This measure primarily assesses the ability to exhale as much air as possible in the shortest amount of time, and is used as an indicator of lung function.

SECONDARY OUTCOMES:
FVC(%predicted), | 52weeks
  FVC (% predicted) was defined as forced vital capacity as a percentage of the predicted value.
FEV1 | 52weeks
  FEV1 (ml/s)was defined as forced expiratory volume in one second.
FEV1 %predicted | 52weeks
  FEV1 (% predicted)was forced expiratory volume in one second as a percentage of the predicted value .
TLC(ml) | 52weeks
  TLC(ml) was defined as Total Lung Capacity.
TLC % predicted | 52weeks
  TLC (% predicted) was defined as total lung capacity as a percentage of the predicted value.
DLco%predicted | 52weeks
  DLco%predicted was diffusing capacity of the lung for carbon monoxide as a percentage of the predicted value.
6-minute walk test | 52weeks
  6-minute walk test is a commonly used method to evaluate physical function and cardiorespiratory health status. The walk distance, usually measured in feet or meters, is an important indicator of the test. It refers to the total distance covered by the subject within 6 minutes, which can reflect their endurance and exercise capacity.
HRCT | 52weeks
  Relative change from baseline in HRCT.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoying Huang, Docter, Principal Investigator — the first affiliated hospital of wenhzou medical university
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- [Background] Raghu G, Collard HR, Egan JJ, Martinez FJ, Behr J, Brown KK, Colby TV, Cordier JF, Flaherty KR, Lasky JA, Lynch DA, Ryu JH, Swigris JJ, Wells AU, Ancochea J, Bouros D, Carvalho C, Costabel U, Ebina M, Hansell DM, Johkoh T, Kim DS, King TE Jr, Kondoh Y, Myers J, Muller NL, Nicholson AG, Richeldi L, Selman M, Dudden RF, Griss BS, Protzko SL, Schunemann HJ; ATS/ERS/JRS/ALAT Committee on Idiopathic Pulmonary Fibrosis. An official ATS/ERS/JRS/ALAT statement: idiopathic pulmonary fibrosis: evidence-based guidelines for diagnosis and management. Am J Respir Crit Care Med. 2011 Mar 15;183(6):788-824. doi: 10.1164/rccm.2009-040GL. PMID 21471066
- [Background] Raghu G. Idiopathic pulmonary fibrosis: lessons from clinical trials over the past 25 years. Eur Respir J. 2017 Oct 26;50(4):1701209. doi: 10.1183/13993003.01209-2017. Print 2017 Oct. PMID 29074545
- [Background] Martinez FJ, Lederer DJ. Focus on Idiopathic Pulmonary Fibrosis: Advancing Approaches to Diagnosis, Prognosis, and Treatment. Chest. 2018 Oct;154(4):978-979. doi: 10.1016/j.chest.2018.08.1021. PMID 30290930
- [Background] Nalysnyk L, Cid-Ruzafa J, Rotella P, Esser D. Incidence and prevalence of idiopathic pulmonary fibrosis: review of the literature. Eur Respir Rev. 2012 Dec 1;21(126):355-61. doi: 10.1183/09059180.00002512. PMID 23204124
- [Background] Raghu G, Remy-Jardin M, Myers JL, Richeldi L, Ryerson CJ, Lederer DJ, Behr J, Cottin V, Danoff SK, Morell F, Flaherty KR, Wells A, Martinez FJ, Azuma A, Bice TJ, Bouros D, Brown KK, Collard HR, Duggal A, Galvin L, Inoue Y, Jenkins RG, Johkoh T, Kazerooni EA, Kitaichi M, Knight SL, Mansour G, Nicholson AG, Pipavath SNJ, Buendia-Roldan I, Selman M, Travis WD, Walsh S, Wilson KC; American Thoracic Society, European Respiratory Society, Japanese Respiratory Society, and Latin American Thoracic Society. Diagnosis of Idiopathic Pulmonary Fibrosis. An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline. Am J Respir Crit Care Med. 2018 Sep 1;198(5):e44-e68. doi: 10.1164/rccm.201807-1255ST. PMID 30168753
- [Background] Lederer DJ, Martinez FJ. Idiopathic Pulmonary Fibrosis. N Engl J Med. 2018 May 10;378(19):1811-1823. doi: 10.1056/NEJMra1705751. No abstract available. PMID 29742380
- [Background] Flaherty KR, Brown KK, Wells AU, Clerisme-Beaty E, Collard HR, Cottin V, Devaraj A, Inoue Y, Le Maulf F, Richeldi L, Schmidt H, Walsh S, Mezzanotte W, Schlenker-Herceg R. Design of the PF-ILD trial: a double-blind, randomised, placebo-controlled phase III trial of nintedanib in patients with progressive fibrosing interstitial lung disease. BMJ Open Respir Res. 2017 Sep 17;4(1):e000212. doi: 10.1136/bmjresp-2017-000212. eCollection 2017. PMID 29018526
- [Background] Wells AU, Brown KK, Flaherty KR, Kolb M, Thannickal VJ; IPF Consensus Working Group. What's in a name? That which we call IPF, by any other name would act the same. Eur Respir J. 2018 May 17;51(5):1800692. doi: 10.1183/13993003.00692-2018. Print 2018 May. PMID 29773608
- [Background] Cottin V, Wollin L, Fischer A, Quaresma M, Stowasser S, Harari S. Fibrosing interstitial lung diseases: knowns and unknowns. Eur Respir Rev. 2019 Feb 27;28(151):180100. doi: 10.1183/16000617.0100-2018. Print 2019 Mar 31. PMID 30814139
- [Background] Kolb M, Vasakova M. The natural history of progressive fibrosing interstitial lung diseases. Respir Res. 2019 Mar 14;20(1):57. doi: 10.1186/s12931-019-1022-1. PMID 30871560
- [Background] Harari S, Caminati A. IPF: new insight on pathogenesis and treatment. Allergy. 2010 May;65(5):537-53. doi: 10.1111/j.1398-9995.2009.02305.x. Epub 2010 Feb 1. PMID 20121758
- [Background] Spagnolo P, Kropski JA, Jones MG, Lee JS, Rossi G, Karampitsakos T, Maher TM, Tzouvelekis A, Ryerson CJ. Idiopathic pulmonary fibrosis: Disease mechanisms and drug development. Pharmacol Ther. 2021 Jun;222:107798. doi: 10.1016/j.pharmthera.2020.107798. Epub 2020 Dec 24. PMID 33359599
- [Background] Richeldi L, du Bois RM, Raghu G, Azuma A, Brown KK, Costabel U, Cottin V, Flaherty KR, Hansell DM, Inoue Y, Kim DS, Kolb M, Nicholson AG, Noble PW, Selman M, Taniguchi H, Brun M, Le Maulf F, Girard M, Stowasser S, Schlenker-Herceg R, Disse B, Collard HR; INPULSIS Trial Investigators. Efficacy and safety of nintedanib in idiopathic pulmonary fibrosis. N Engl J Med. 2014 May 29;370(22):2071-82. doi: 10.1056/NEJMoa1402584. Epub 2014 May 18. PMID 24836310
- [Background] Richeldi L, Kreuter M, Selman M, Crestani B, Kirsten AM, Wuyts WA, Xu Z, Bernois K, Stowasser S, Quaresma M, Costabel U. Long-term treatment of patients with idiopathic pulmonary fibrosis with nintedanib: results from the TOMORROW trial and its open-label extension. Thorax. 2018 Jun;73(6):581-583. doi: 10.1136/thoraxjnl-2016-209701. Epub 2017 Oct 9. PMID 28993537
- [Background] Noble PW, Albera C, Bradford WZ, Costabel U, Glassberg MK, Kardatzke D, King TE Jr, Lancaster L, Sahn SA, Szwarcberg J, Valeyre D, du Bois RM; CAPACITY Study Group. Pirfenidone in patients with idiopathic pulmonary fibrosis (CAPACITY): two randomised trials. Lancet. 2011 May 21;377(9779):1760-9. doi: 10.1016/S0140-6736(11)60405-4. Epub 2011 May 13. PMID 21571362
- [Background] King TE Jr, Bradford WZ, Castro-Bernardini S, Fagan EA, Glaspole I, Glassberg MK, Gorina E, Hopkins PM, Kardatzke D, Lancaster L, Lederer DJ, Nathan SD, Pereira CA, Sahn SA, Sussman R, Swigris JJ, Noble PW; ASCEND Study Group. A phase 3 trial of pirfenidone in patients with idiopathic pulmonary fibrosis. N Engl J Med. 2014 May 29;370(22):2083-92. doi: 10.1056/NEJMoa1402582. Epub 2014 May 18. PMID 24836312
- [Background] Costabel U, Albera C, Glassberg MK, Lancaster LH, Wuyts WA, Petzinger U, Gilberg F, Kirchgaessler KU, Noble PW. Effect of pirfenidone in patients with more advanced idiopathic pulmonary fibrosis. Respir Res. 2019 Mar 12;20(1):55. doi: 10.1186/s12931-019-1021-2. PMID 30866942
- [Background] Ruan H, Lv Z, Liu S, Zhang L, Huang K, Gao S, Gan W, Liu X, Zhang S, Helian K, Li X, Zhou H, Yang C. Anlotinib attenuated bleomycin-induced pulmonary fibrosis via the TGF-beta1 signalling pathway. J Pharm Pharmacol. 2020 Jan;72(1):44-55. doi: 10.1111/jphp.13183. Epub 2019 Oct 28. PMID 31659758
- [Background] Nair AB, Jacob S. A simple practice guide for dose conversion between animals and human. J Basic Clin Pharm. 2016 Mar;7(2):27-31. doi: 10.4103/0976-0105.177703. PMID 27057123